CLINICAL TRIAL: NCT06543420
Title: The Role of Levator Ani Muscle Reconstruction Technology in Urinary Incontinence Recovery After Robot Assisted Radical Prostatectomy: a Randomized Controlled Clinical Trial
Brief Title: The Role of Levator Ani Muscle Reconstruction Technology in Urinary Incontinence Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, GONG Kan, Chief physician, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chfcj2024
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Levator ani muscle reconstruction; Urinary incontinence recovery; Robot-assisted radical prostatectomy; Randomized controlled trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Posterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lateral reconstruction group (Experimental): After RARP surgery, lateral reconstruction is performed
  Interventions: Procedure: lateral reconstruction
- posterior reconstruction group (Experimental): After RARP surgery, posterior reconstruction is performed
  Interventions: Procedure: posterior reconstruction
- control group (No Intervention): No lateral or posterior reconstruction is performed after RARP surgery

INTERVENTIONS:
Procedure: lateral reconstruction — In lateral reconstruction group, lateral reconstruction is performed by suturing the levator ani muscle to the prostatic collateral ligament and fascia to strengthen the lateral posterior support structure.
  Arms: lateral reconstruction group
Procedure: posterior reconstruction — In posterior group, prior to completion of the operation, the posterior fibrous tissues of the sphincter are joined to the residual Denonvilliers fascia on the posterior bladder wall 1-2 cm cephalad and dorsally to the new bladder neck.
  Arms: posterior reconstruction group

SUMMARY:
This study is a single center, single blind, prospective randomized controlled trial. Patients undergoing robot assisted laparoscopic radical prostatectomy for prostate cancer were randomly divided into 1:1:1 groups, using lateral reconstruction, posterior reconstruction, or no reconstruction. Patients were followed up regularly after surgery and clinical data were collected, including daily use of urine pads, ICIQ-SF score, 24-hour urine leakage, I-QoL score, etc., to evaluate the improvement effect of lateral reconstruction on urinary control and the difference in effect between lateral reconstruction and posterior reconstruction, thereby improving the quality of life of prostate cancer patients after surgery.

DETAILED DESCRIPTION:
This study is a single center, single blind, prospective randomized controlled trial. Collect baseline data from enrolled patients Materials were randomly divided into experimental group A (lateral reconstruction group), experimental group B (posterior reconstruction group), and control group (non reconstruction group) in a 1:1:1 ratio using a computer-generated random number sequence.

In the control group (non reconstruction group), no lateral or posterior reconstruction was performed after RARP surgery.

In experimental group A (lateral reconstruction group), lateral reconstruction was performed after RARP surgery, in which the levator ani muscle was sutured to the prostatic collateral ligament and fascia to strengthen the lateral posterior support structure.

In experimental group B (post reconstruction group), post reconstruction was performed after RARP surgery.

This study used blinding on patients to avoid subjective factors affecting the results of whether reconstruction was performed or not.

Preoperative collection of baseline data from patients includes age, BMI, history of abdominal surgery, most recent PSA, PI-RADS score, prostate volume, prostate puncture related data (histological type, number of positive needles/puncture needles, Gleason score, maximum tumor proportion), PSMA PET-CT results, neoadjuvant therapy regimen, International Advisory Committee on Urinary Incontinence Questionnaire Brief (ICIQ-SF) score, International Index of Erectile Function (IIEF-5) score, International Prostate Symptom Score (IPSS) score, etc.

Collect postoperative patient surgical data (including ASA score, surgical duration, intraoperative blood loss, etc.), hospitalization data (including hospitalization duration, hospitalization costs, etc.), and pathological data (including lesion diameter, histological type, Gleason score, pathological staging, positive surgical margin, invasion of capsule, invasion of seminal vesicle and adjacent tissues, etc.).

Follow up visits were conducted on patients at 1, 3, 6, 9, and 12 months postoperatively, and relevant clinical data were collected, including the number of urine pads used per day during follow-up, ICIQ-SF score, 24-hour urine leakage (accurately measured by purchasing an electronic scale for patients), perioperative and postoperative complications, IIEF-5 score, PSA, and urinary incontinence quality of life questionnaire (I-QOL) score, in order to evaluate the improvement effect of lateral reconstruction on urinary control and quality of life, as well as the impact on complication incidence, erectile function, and tumor control. The differences in the effects of lateral reconstruction and posterior reconstruction on urinary control recovery and quality of life improvement were compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer and preoperative clinical stage of cT2~T3aN0M0
* Complies with the indications for RARP surgery

Exclusion Criteria:

* History of urinary incontinence or urethral stricture
* Previous prostate related surgical treatment
* Contraindications for RARP surgery
* The patient or their family members refuse to participate

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of urinary incontinence | 1,3,6,9,12 months after operation
  Urinary incontinence recovery is defined as using 0 urinary pads per day

SECONDARY OUTCOMES:
The International Consultation on Incontinence Questionnaire Short-form(ICIQ-SF) Score | 1,3,6,9,12 months after operation
  ICIQ-SF is a questionnaire used to evaluate urinary incontinence and assess the recovery of postoperative urinary incontinence in patients. The range of scores is from 0 to 21, with higher scores indicating more severe urinary incontinence.
Incontinence Quality of Life Questionnaire(I-QOL) Score | 1,3,6,9,12 months after operation
  I-QoL is a questionnaire used to evaluate the quality of life of patients with urinary incontinence after surgery. The range of scores is from 0 to 100, with higher scores indicating higher quality of life.
Perioperative and postoperative complications | 1,3,6,9,12 months after operation
  Collect perioperative and postoperative complications such as bleeding and pain to compare the differences between two reconstruction methods and non reconstruction methods.
Prostate-specific antigen | 1,3,6,9,12 months after operation
  Biochemical recurrence is defined as two consecutive postoperative PSA levels above 0.2 ng/ml with an upward trend
Duration of operation | immediately after operation
  The purpose of collecting surgical duration is to compare whether there are differences between two reconstruction techniques and no reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China